CLINICAL TRIAL: NCT05426525
Title: Use of Empagliflozin to Treat Prediabetes - a Randomized, Double-blind, Placebo-controlled 13-week Intervention Trial
Brief Title: Use of Empagliflozin to Treat Prediabetes
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Samaritan Health Services (Other)
Responsible Party: Principal Investigator, Sean Newsom, Associate Professor, Kinesiology, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OregonSU
Record Dates: First submitted 2022-06-08; First posted 2022-06-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: PreDiabetes; Prediabetic State; Overweight and Obesity
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pills will be prepared and dispensed by a pharmacy to blind participants and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Participants will be provided 10-25mg empagliflozin per day for 13 weeks.
  Interventions: Drug: Empagliflozin
- Multivitamin-Placebo (Placebo Comparator): Participants will be provided 1 multivitamin-placebo per day for 13 weeks.
  Interventions: Drug: Multivitamin-Placebo

INTERVENTIONS:
Drug: Empagliflozin — Participants will take 10mg empagliflozin per day for 2 weeks. Absent contraindications, dosing will be increased to 25 mg empagliflozin per day for the next 11 weeks.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Multivitamin-Placebo — Participants will take 1 multivitamin per day for 13 weeks.
  Arms: Multivitamin-Placebo

SUMMARY:
The overall purpose of this study is to identify how empagliflozin (a drug commonly used to treat type 2 diabetes) impacts skeletal muscle metabolic health among adults with prediabetes. Our aims are to: 1) Test the ability of empagliflozin to improve regulation of glucose metabolism (i.e., blood sugar) among overweight and obese individuals at risk for diabetes, and 2) Identify mechanisms to explain how empagliflozin may improve skeletal muscle glucose metabolism. We hypothesize empagliflozin will improve regulation of glucose metabolism due to changes in whole-body and skeletal muscle metabolism (e.g., increased rates of whole-body fat oxidation, evidence of impaired skeletal muscle mitochondrial respiratory function and increased energetic stress, lower accumulation of skeletal muscle lipids and improved skeletal muscle insulin signaling compared with placebo treatment).

DETAILED DESCRIPTION:
The overall study design is a 13-week, double-blind, placebo-controlled intervention trial, testing the ability of empagliflozin to improve glucose metabolism among overweight and obese individuals at risk for diabetes (compared with a multivitamin-placebo). The study involves metabolic testing before and during the intervention to identify changes in outcomes as a function of the intervention and to ensure participant safety. The study involves 9 visits to the Samaritan Athletic Medicine Center on the campus of Oregon State University in Corvallis, Oregon. Full completion of the study is anticipated to take ~4 months. The project is being completed in collaboration with physicians at Samaritan Health Services.

ELIGIBILITY:
Inclusion Criteria:

* BMI 26-45 kg/m2
* Weight stable (± 10 lbs in previous 3 months)
* Fasting blood glucose <126 mg/dL or HbA1c <6.5% (<48mmol/mol)

Exclusion Criteria:

* Regular moderate-vigorous exercise (≥30 min/session on ≥2 days per week)
* Pregnancy, planning to become pregnant or nursing
* Lidocaine allergy
* Current or recent smoking or nicotine use (≤ 1-year abstention)
* Medications including glucose lowering medications and supplements (SGLT2 inhibitors, GLP1 agonists, sulfonylurea, insulin, TZDs); mono-amine oxidase inhibitors; beta-blockers; diuretics
* Major metabolic or cardiovascular conditions (e.g., type 1 diabetes, Crohn's disease, untreated hypo- or hyperthyroid, cancer, coronary artery disease, tachycardia, prior bariatric surgery, peripheral vascular disease, liver diseases (e.g., cirrhosis)
* Diagnosed type 2 diabetes. In absence of diagnosis, two separate samples with test results of fasting blood glucose ≥126 mg/dL or HbA1c ≥6.5% (48 mmol/mol).
* Contraindications/precautions for empagliflozin (impaired renal function (EGR<60), history of: empagliflozin hypersensitivity, ketoacidosis, hypotension, recurring urinary tract or genital mycotic infections, amputation)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Insulin-stimulated glucose disposal | Insulin-stimulated glucose disposal is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  The glucose infusion rate to maintain glycemia during insulin clamp, using plasma enrichment of glucose isotope tracer to determine changes in rates of insulin-stimulated glucose disposal

SECONDARY OUTCOMES:
Oral glucose tolerance | Oral glucose tolerance is measured before the start of the intervention (baseline) and during week 12 of the intervention.
  The change in blood glucose concentration in response to a 75g glucose beverage
Fasting plasma glucose concentration | Fasting plasma glucose is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  The change in fasting plasma glucose concentration
Whole-body fat oxidation | Whole-body fat oxidation is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  Indirect calorimetry will be used to determine the change in whole-body rate of fat oxidation during basal and insulin-stimulated conditions
Skeletal muscle insulin signaling | Skeletal muscle insulin signaling is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  Immunoblotting to determine the change in activation of insulin signaling proteins in skeletal muscle collected at basal and during insulin-stimulated conditions
Skeletal muscle lipids | Skeletal muscle lipids are measured before the start of the intervention (baseline) and during week 13 of the intervention.
  Mass spectrometry lipidomic analysis of skeletal muscle to determine changes in muscle lipid content
Skeletal muscle mitochondrial respiratory function | Skeletal muscle mitochondrial respiratory function is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  Changes in skeletal muscle mitochondrial respiratory capacity measured using high-resolution respirometry
Skeletal muscle energetic stress | Skeletal muscle energetic stress is measured before the start of the intervention (baseline) and during week 13 of the intervention.
  Immunoblotting to determine changes in activation of AMPK and related signaling proteins pathways

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Newsom, Ph.D., Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The current study is a pilot and feasibility project. IPD will not be made publicly available, save for publication and reporting requirements. Individual requests for data will be addressed by the Principal Investigator.